CLINICAL TRIAL: NCT05434390
Title: Evaluating the Feasibility and Acceptability of a Latino MSM Focused PrEP Uptake Intervention
Brief Title: A Latino MSM Focused Pre-Exposure Prophylaxis Uptake Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bienestar Human Services, Inc. (Other)
Responsible Party: Principal Investigator, Ronald Andrew Brooks, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#21-002132
Record Dates: First submitted 2022-06-09; First posted 2022-06-28 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-06

CONDITIONS: HIV
Keywords: HIV prevention; Pre-exposure prophylaxis; Latino men who have sex with men

STUDY DESIGN:
Intervention Model Description: Parallel model. Participants will be randomly assigned to either an intervention or control arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latino MSM PrEP intervention (Experimental): The Latino MSM PrEP intervention consists of 4 small group sessions with concurrent peer navigation and counseling.
  Interventions: Behavioral: Estoy PrEParado/ I am PrEPared intervention
- Control condition (Active Comparator): The control condition consists of usual care at the study site (i.e., referrals to PrEP services).
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Estoy PrEParado/ I am PrEPared intervention — Participants will receive an Information, Motivation, and Behavioral skills model PrEP intervention tailored for mixed immigrant status Latino men who have sex with men
  Arms: Latino MSM PrEP intervention
Behavioral: Usual Care — Participants will be offered PrEP navigation services as part of usual care at the study site.
  Arms: Control condition

SUMMARY:
The clinical study will evaluate the feasibility and acceptability of a culturally tailored behavioral intervention to improve uptake of pre-exposure prophylaxis for HIV prevention among at-risk Latino men who have sex with men.

DETAILED DESCRIPTION:
The clinical study will evaluate the feasibility and acceptability of a brief small group and peer navigation behavioral intervention to improve uptake of pre-exposure prophylaxis (PrEP) for HIV prevention among at-risk Latino men who have sex with men. The brief intervention consists of 4 small group sessions with concurrent peer navigation and counseling. Study participants will be randomized to either an intervention or control condition. Participants in the control condition will receive usual care for PrEP promotion (i.e., referral to PrEP services). The study will determine the feasibility and acceptability of the intervention among Latino men who have sex with men and assess the preliminary impact of the intervention compared to control condition in facilitating PrEP uptake.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* assigned male at birth
* Identifies as Latino/Hispanic origin
* HIV-negative or HIV status unknown
* Man who has had sex with other men in the past 24 months
* Not currently using PrEP for HIV prevention

Exclusion Criteria:

* Male under 18 years of age
* Not identifying as being of Latino/Hispanic origin
* Man who has not had sex with other men in the past 24 months
* Identifies as cisgender or transgender Female/woman
* Assigned female at birth

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender male
Enrollment: 80 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | assessed at 1-month follow-up
  We will assess PrEP uptake using evidence of a prescription for Truvada® or Descovy® (participant shows us their prescription bottle in person or via a text photo).
PrEP initiation | assessed at 3-month follow-up
  We will assess PrEP uptake using evidence of a prescription for Truvada® or Descovy® (participant shows us their prescription bottle in person or via a text photo).
PrEP adherence single measure | assessed at 1-month follow-up
  We will assess adherence to the PrEP medication using a single-item self-rating adherence measure.
PrEP adherence single measure | assessed at 3-month follow-up
  We will assess adherence to the PrEP medication using a single-item self-rating adherence measure.
PrEP adherence urine sample | assessed at 1-month follow-up
  We will assess adherence to the PrEP medication by analyzing participants' urine sample to determine the presence of the medication tenofovir, a key medication in the PrEP medication.
PrEP adherence urine sample | assessed at 3-month follow-up
  We will assess adherence to the PrEP medication by analyzing participants' urine sample to determine the presence of the medication tenofovir, a key medication in the PrEP medication.

SECONDARY OUTCOMES:
Changes in Readiness to Adopt PrEP | assessed at 1-month follow-up
  We will assess changes in readiness to adopt PrEP using the PrEP Transtheoretical Stages of Change Model measure (pre-contemplation, contemplation, preparation, action & initiation, and maintenance).
Changes in Readiness to Adopt PrEP | assessed at 3-month follow-up
  We will assess changes in readiness to adopt PrEP using the PrEP Transtheoretical Stages of Change Model measure (pre-contemplation, contemplation, preparation, action & initiation, and maintenance).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald A Brooks, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Bienestar Human Services, Los Angeles, California, United States